CLINICAL TRIAL: NCT00631839
Title: Prospect Study to Evaluate Clinical, Dosimetrical, Functional, Biological and Genetic Factors in Predicting Chemo-Radiotherapy Induced Lung and Esophagus Injury
Brief Title: Prospective Study on Factors Predicting Chemo-Radiotherapy Induced Pulmonary and Esophageal Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Fan Min, Associate Professor, Vice Chief of Lung Cancer Center, Fudan University, Shanghai Cancer Hospital, China
Other Study IDs: FDCA002
Record Dates: First submitted 2008-03-02; First posted 2008-03-10 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Thoracic Neoplasms
Keywords: Thoracic Neoplasms; Platinum-based chemotherapy; 3-D Conformal Radiotherapy; Chemo-radiotherapy induced lung injury; Chemo-radiotherapy induced esophagus injury
MeSH Terms: conditions — Thoracic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients' blood samples will be retained for the purpose of cytokine and MnSOD assay and DNA detection. The samples will be left till the study ends. Paitents will have their vein blood drawn from left arm 6am every Monday during RT. All above is stated in informed consent form.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: There is only one group in this study. The patients of this group will go through procedures as follow: basic pre-treatment information collected,treatment include platinum-based chemotherapy and 3-D conformal radiotherapy, blood test during RT 6am every Monday and follow-up visits with treatment-induced injury assessed.
  Interventions: Radiation: Thoracic 3-D Conformal Radiotherapy

INTERVENTIONS:
Radiation: Thoracic 3-D Conformal Radiotherapy — Thoracic RT tailored for each patient, about 60Gy (NSCLC) or 55Gy (SCLC) with photon energies >=6MV.
  Other Names: Thoracic Radiotherapy(TRT)

SUMMARY:
The purpose of this study is to evaluate clinical, dosimetrical, functional, biological and genetic factors in predicting chemo-radiotherapy induced lung and esophagus injury.

DETAILED DESCRIPTION:
We propose a prospective study to investigate the combinational effect of radiotherapeutic dosimetric parameters [mean lung dose and percentage of lung volume receiving at least XGy (Vx)] and biological parameters [interleukin-1α(IL1α),interleukin-1β(IL1β),interleukin-6(IL6),interleukin-7(IL7),transforming growth factor beta (TGFB)] and manganese superoxide dismutase(MnSOD) in predicting radiation pneumonitis, fibrosis, and radiation esophageal injury. Eligibility included pathological or cytological proven thoracic cancer,ECOG performance status [PS] 0-2, no prior thoracic RT or chemotherapy,no distant metastasis and signed informed consent prior to study entry.

Basic pre-treatment information will be collected, which included ECOG PS, UICC/AJCC stage,primary lesion site, history of smoking/coexisting lung disease/surgical resection, and pulmonary function test of FEV1/VC/DLCO. Computed tomography [CT] of the whole lung in treatment position. Blood test of IL1α,IL1β,IL6,IL7,TGFB and MnSOD by ELISA will be done before and weekly during RT. RT must be given by photon energies >=6MV. Radiation lung and esophageal injury will be assessed according to common toxicity criteria adverse effect version3.0 [CTCAE-3.0] during RT and in every follow up visits. Genomic DNA is obtained from the blood drawn during RT. Chi-square test, T test, analysis of variance, logistic regression, and proportional hazard ratio method will be used to investigate whether the parameter(s) can be effective in predicting radiation related sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adults (18<= age <= 75 y/o)
* Chinese ethnicity
* Pathological or cytological proven thoracic neoplasms (of note,sputum cytology alone is not acceptable.Cytological specimens obtained by brushing,washing and needle aspiration of a defined lesion are acceptable)
* Initially treated
* No distant metastasis
* ECOG PS 0-2 (Karnofsky>60%)
* Understand and willing to sign the consent
* Normal organ and marrow function as defined below:

  * Leukocytes >=3,000/µL
  * Haemoglobin >=9 g/dL (prior to transfusions)
  * Absolute neutrophil count >=1,500/µL
  * Platelets >=100,000/µL
  * Total bilirubin < 1.5 x upper limit of normal
  * AST (SGOT)/ALT (SGPT) ≤2.5 X institutional upper limit of normal
  * Creatinine <=2.5 mg/dl.

Exclusion Criteria:

* Prior thoracic radiotherapy
* Distant metastasis
* Allergic reactions attributed to compounds of similar chemical or biologic composition to platinum-based drugs.
* Pre-existed non-oncological pulmonary or esophageal disease that may put the patient at high risk of severe toxicities.
* Other uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would limit compliance with study requirement
* pregnancy or lactating
* Receiving other investigational agents or devices

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled are Chinese with thoracic neoplasms, no distant metastasis and initially treated.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2002-01; Primary Completion 2006-01 (Actual); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Chemo-Radiotherapy induced pneumonitis,fibrosis and esophagus injury assessed with common toxicity criteria adverse effect version3.0 [CTCAE-3.0] | from the begining of treatment to the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Min Fan, MD, Principal Investigator — Fudan University Cancer Hospital, Department of Radiation Oncology
Locations (1):
- Fudan University, Cancer Hospital, Department of Radiation Oncology, Shanghai, China